CLINICAL TRIAL: NCT02549664
Title: Exercise in Genetic Cardiovascular Conditions (Lifestyle and Exercise in Hypertrophic Cardiomyopathy "LIVE-HCM"/Lifestyle and Exercise in the Long QT Syndrome "LIVE-LQTS"
Brief Title: Exercise in Genetic Cardiovascular Conditions
Acronym: LIVE-HCM/LQT
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1411014982; 1R01HL125918-01 (NIH)
Record Dates: First submitted 2015-06-10; First posted 2015-09-15 (Estimated); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Hypertrophic Cardiomyopathy; Long QT Syndrome
Keywords: Hypertrophic Cardiomyopathy (HCM); Long QT Syndrome (LQTS)
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Long QT Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- LQT/HCM sedentary patients: LQT/HCM sedentary lifestyle
- LQT/HCM moderate/vigorous exercise: LQT/HCM participate in moderate or vigorous exercise

SUMMARY:
The goal is to determine how lifestyle and exercise impact the well-being of individuals with hypertrophic cardiomyopathy (HCM) and long QT syndrome (LQTS).

Ancillary study Aim: To understand how the coronavirus epidemic is impacting psychological health and quality of life in the LIVE population

DETAILED DESCRIPTION:
Yale is the central site for this multicenter study. Patients with HCM and LQTS will be recruited via high-volume HCM and LQTS sites, patient-groups, and websites. Information about exercise participation will be acquired via interview and online instruments at enrollment and every six months for three years. Quality of Life questionnaires will be filled out at enrollment and at the end of the study. Participants will receive a Fitbit (pedometer) and will wear it initially for two weeks and then one week every three months. The Fitbit is used for assessment of exercise level only. Clinical records will be obtained from treating physicians. Participants will also be asked to call the central site if they experience syncope, appropriate ICD (implantable cardioverter defibrillator) shock, or resuscitated arrest. Information regarding the patient's activity at the time of event will then be obtained by phone interview. Follow-up clinical records will be obtained as indicated to corroborate endpoints.

The Ancillary study is optional. This will include all of the baseline questionnaires,as well as selected questions from the Epi-Pandemic Impacts Inventory.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with Hypertrophic Cardiomyopathy or Long QT Syndrome

Exclusion Criteria:

* Individuals with Hypertrophic Cardiomyopathy with systolic or diastolic heart failure which precludes vigorous exercise will not be enrolled (NYHA III/IV)

Ages: 8 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Individuals with Hypertrophic Cardiomyopathy or Long QT Syndrome between the ages of 8-60.
Sampling Method: Non-Probability Sample
Enrollment: 4299 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
To compare composite risk of death, cardiac arrest, ventricular arrhythmias, or syncope in individuals with HCM or LQTS who are participating in moderate or vigorous exercise and in sedentary individuals. | Five years
  Collect information for death, resuscitated arrest, syncope, appropriate ICD shock , during exercise or at other times, through records from the provider and patient interviews

SECONDARY OUTCOMES:
Emotional Quality of Life assessed using Pediatric Cardiac Quality of Life Inventory (Pcqli) | Five years
  Will assess using Pediatric Cardiac Quality of Life Inventory (Pcqli)
Physical Quality of Life assessed using Pediatric Quality of Life Inventory (PedsQL) | Five Years
  Will assess using Pediatric Quality of Life Inventory (PedsQL)
Physical Quality of Life assessed using Health Status Questionnaire (SF36) Quality of Life for Adults | Five Years
  Will assess using Health Status Questionnaire (SF36) Quality of Life for Adults

OTHER OUTCOMES:
Epi-Pandemic Impacts Inventory (select questions) | 4 months
  Will assess COVID 19 infection in themselves/family/friends, and impact on jobs and financial status.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Lampert, MD, Principal Investigator — Yale University
Locations (36):
- United States (29):
  - University of Arizona, Tucson, Arizona
  - University of California Irvine, Orange, California
  - University of California, San Diego (Rady's Children's Hospital), San Diego, California
  - Stanford, Stanford, California
  - Yale University, New Haven, Connecticut
  - Children's National, Washington D.C., District of Columbia
  - Miami Children's (Nicklaus Children's Hospital), Miami, Florida
  - Lurie Children's, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Louisville, Louisville, Kentucky
  - Johns Hopkins, Baltimore, Maryland
  - Tufts, Boston, Massachusetts
  - Boston Children's, Boston, Massachusetts
  - Brigham & Women's, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Children's Omaha, Omaha, Nebraska
  - NYU, New York, New York
  - Cincinnati Children's, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science, Portland, Oregon
  - Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - UT Southwestern, Dallas, Texas
  - Texas Children's, Houston, Texas
  - University of Utah (Primary Children's), Salt Lake City, Utah
  - Seattle Children's, Seattle, Washington
- Royal Prince Alfred Hospital/Sydney AU, Camperdown, New South Wales, Australia
- Canada (3):
  - University of BC, Providence Health, Vancouver, British Columbia
  - University of BC, Children's, Vancouver, British Columbia
  - University of Toronto, Toronto, Ontario
- Starship Children's Hospital, Grafton, Auckland, New Zealand
- United Kingdom (2):
  - St. Georges, London, London, England
  - Royal Brompton Hospital, London, England

REFERENCES:
- [Derived] Lampert R, Day S, Ainsworth B, Burg M, Marino BS, Salberg L, Tome Esteban MT, Abrams DJ, Aziz PF, Barth C, Behr ER, Bell C, Berul CI, Bos JM, Bradley D, Cannom DS, Cannon BC, Concannon MA, Cerrone M, Czosek RJ, Dubin AM, Dziura J, Erickson CC, Estes NAM 3rd, Etheridge SP, Goldenberg I, Gray B, Haglund-Turnquist C, Harmon K, James CA, Johnsrude C, Kannankeril P, Lara A, Law IH, Li F, Link MS, Molossi SM, Olshansky B, Noseworthy PA, Saarel EV, Sanatani S, Shah M, Simone L, Skinner J, Tomaselli GF, Ware JS, Webster G, Zareba W, Zipes DP, Ackerman MJ. Vigorous Exercise in Patients With Congenital Long QT Syndrome: Results of the Prospective, Observational, Multinational LIVE-LQTS Study. Circulation. 2024 Aug 13;150(7):516-530. doi: 10.1161/CIRCULATIONAHA.123.067590. Epub 2024 Jul 25. PMID 39051104
- [Derived] Lee TM, Hsu DT, Kantor P, Towbin JA, Ware SM, Colan SD, Chung WK, Jefferies JL, Rossano JW, Castleberry CD, Addonizio LJ, Lal AK, Lamour JM, Miller EM, Thrush PT, Czachor JD, Razoky H, Hill A, Lipshultz SE. Pediatric Cardiomyopathies. Circ Res. 2017 Sep 15;121(7):855-873. doi: 10.1161/CIRCRESAHA.116.309386. PMID 28912187